CLINICAL TRIAL: NCT06726148
Title: An Open-label, Multi-center, Phase I/II Study of ECI830 as a Single Agent and in Combination With Ribociclib and Endocrine Therapy in Patients With Advanced Hormone Receptor Positive, HER2-negative Breast Cancer and Advanced Solid Tumors
Brief Title: Study of ECI830 Single Agent or in Combination in Patients With Advanced HR+/HER2- Breast Cancer and Other Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CECI830A12101; 2024-517281-42 (Registry Identifier: CTIS)
Expanded Access: NCT05038631 (Available)
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Advanced HR+/HER2- Breast Cancer; Advanced CCNE1-amplified Solid Tumors
Keywords: ECI830; Ribociclib; Fulvestrant; Breast cancer; CCNE1 amplification
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- ECI830 Single Agent (Arm A) (Experimental): Phase I
  Interventions: Drug: ECI830
- Dose Escalation Combination ECI830 + ribociclib + fulvestrant (Arm B) (Experimental): Phase I
  Interventions: Drug: ECI830; Drug: ribociclib; Drug: fulvestrant
- Ribociclib in combination with fulvestrant (Arm C) (Experimental): Phase II
  Interventions: Drug: ribociclib; Drug: fulvestrant
- ECI830 in combination with fulvestrant (Arm D) (Experimental): Phase II
  Interventions: Drug: ECI830; Drug: fulvestrant
- ECI830 in combination with ribociclib and fulvestrant (Arm E) (Experimental): Phase II
  Interventions: Drug: ECI830; Drug: ribociclib; Drug: fulvestrant
- ECI830 in combination with ribociclib and fulvestrant (Arm F) (Experimental): Phase II
  Interventions: Drug: ECI830; Drug: ribociclib; Drug: fulvestrant

INTERVENTIONS:
Drug: ECI830 — Experimental
  Arms: Dose Escalation Combination ECI830 + ribociclib + fulvestrant (Arm B); ECI830 Single Agent (Arm A); ECI830 in combination with fulvestrant (Arm D); ECI830 in combination with ribociclib and fulvestrant (Arm E); ECI830 in combination with ribociclib and fulvestrant (Arm F)
Drug: ribociclib — Approved medication
  Other Names: Kisqali
  Arms: Dose Escalation Combination ECI830 + ribociclib + fulvestrant (Arm B); ECI830 in combination with ribociclib and fulvestrant (Arm E); ECI830 in combination with ribociclib and fulvestrant (Arm F); Ribociclib in combination with fulvestrant (Arm C)
Drug: fulvestrant — Approved medication
  Other Names: Faslodex
  Arms: Dose Escalation Combination ECI830 + ribociclib + fulvestrant (Arm B); ECI830 in combination with fulvestrant (Arm D); ECI830 in combination with ribociclib and fulvestrant (Arm E); ECI830 in combination with ribociclib and fulvestrant (Arm F); Ribociclib in combination with fulvestrant (Arm C)

SUMMARY:
Phase I: Characterize safety and tolerability of ECI830 as a single agent and in combination with ribociclib and fulvestrant. Identify dose range for optimization/recommended dose for future studies.

Phase II: Assess the anti-tumor activity of ECI830 in combination with ribociclib and fulvestrant in patients with hormone receptor-positive/human epidermal growth factor receptor 2-negative (HR+/HER2-) advanced breast cancer.

DETAILED DESCRIPTION:
This is a first-in-human, open-label, phase I/II, multi-center study consisting of an ECI830 single agent treatment arm in patients with advanced HR+/HER2- breast cancer or other advanced solid tumors harboring CCNE1 amplification and a combination treatment arm of ECI830 with ribociclib and fulvestrant in patients with advanced breast cancer. Single agent escalation may be followed by an expansion part stratified by disease indication. The escalation of the combination arm may continue into a randomized, open label, Phase II with optional dose optimization in advanced breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years old.

Patients with one of the following indications:

Phase I:

HR+/HER2- aBC with disease progression on or following at least one line of hormone-based therapy in combination with a CDK4/6i and at least one additional line of systemic therapy for metastatic disease.

Histologically and/or cytologically confirmed diagnosis of locally advanced or metastatic cancer with a CCNE1 amplification. For dose expansion only: no more than 3 prior lines of therapy for advanced or metastatic disease.

Phase II:

HR+/HER2- aBC with disease progression on an aromatase inhibitor or tamoxifen in combination with a CDK4/6 inhibitor for unresectable/metastatic disease with no more than 2 lines of endocrine therapy.

Measurable disease as determined by RECIST v1.1.

BC only: If no measurable disease is present, then at least one predominantly lytic bone lesion must be present that can be accurately assessed at baseline and is suitable for repeated assessment.

Exclusion Criteria:

Previous treatment with a CDK2 inhibitor at any time.

Patients with inadequate bone marrow and/or organ functions with out-of-range laboratory values.

Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality including MI, CABG, long QT syndrome, or risk factors for TdP.

Presence of symptomatic CNS metastases or CNS metastases that require local therapy or increasing doses of corticosteroids within 2 weeks prior to study entry.

For the combination treatment:

Patients with symptomatic visceral disease or any disease burden that makes the patient ineligible for endocrine-based therapy.

Patients who could not tolerate the prescribed dose of ribociclib during a previous course of treatment, requiring dose reduction or permanent discontinuation due to adverse events.

For patients with BC: Patient is concurrently using hormone replacement therapy.

WOCBP who are unwilling to use highly effective contraception methods, pregnant or nursing women.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2028-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of dose-limiting toxicities (DLTs) | 2 years
  A DLT is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications that occurs within the first 28 days of treatment. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Phase I: Incidence of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Number of participants with AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Phase I: Number of participants with dose interruptions, reductions and discontinuations | 2 years
  Assessment of tolerability. For patients who do not tolerate the protocol-specified dosing schedule, dose adjustments are permitted in order to allow patients to continue the study treatment.
Phase II: PFS rate at 6 months per local response evaluation criteria in solid tumors (RECIST) v1.1 | 6 months
  Progression Free Survival (PFS) rate at 6 months is defined as the proportion of patients who are alive and progression-free per RECIST v1.1 at 6 months.

SECONDARY OUTCOMES:
Phase I and II: Area under the plasma concentration-time curve (AUC) of ECI830 and ribociclib | From pre-dose up to 24 hours post-dose in Cycle 1. One cycle=28 days.
  Pharmacokinetic (PK) parameters calculated based on ECI830 and ribociclib plasma concentrations by using non-compartmental methods.
Phase I and II: Maximum observed plasma concentration (Cmax) of ECI830 and ribociclib | From pre-dose up to 24 hours post-dose in Cycle 1. One cycle=28 days.
  PK parameters calculated based on ECI830 and ribociclib plasma concentrations by using non-compartmental methods.
Phase I and II: Best overall response (BOR) per RECIST v1.1 | 2 years
  BOR per RECIST v1.1 is defined as the best overall confirmed response recorded from the start of the treatment until progressive disease (PD), death, start of new therapy, withdrawal of consent or end of study, whatever comes first.
Phase I and II: Overall response rate (ORR) per RECIST v1.1 | 2 years
  ORR per RECIST v1.1 is defined as the proportion of patients with a BOR of Complete response (CR) or Partial response (PR) according to RECIST v1.1 as per local review.
Phase I and II: Disease control rate (DCR) per RECIST v1.1 | 2 years
  DCR per RECIST v1.1 is defined as the proportion of patients with a BOR of CR, PR, or Stable disease (SD) according to RECIST v1.1 as per local review.
Phase I and II: Clinical benefit rate (CBR) per RECIST v1.1 | 2 years
  CBR per RECIST v1.1 is defined as the proportion of patients with a BOR of CR, PR, or an overall lesion response of SD or Non-CR/Non-PD which lasts for at least 24 weeks according to RECIST v1.1 as per local review.
Phase I and II: Progression Free Survival (PFS) per RECIST v1.1 | 2 years
  PFS is defined as the time from the date randomization to the date of the first documented progression or death due to any cause.
Phase II: Duration of Response (DOR) per RECIST v1.1 | 2 years
  DOR per RECIST v1.1 is the time between the first documented response (CR or PR) and the date of progression or death due to any cause.
Phase II: Overall Survival (OS) | 2 years
  OS is defined as the time between the date of randomization to the date of death due to any cause.
Phase II: Incidence of adverse events (AEs) and serious adverse events (SAEs) | 2 years
  Number of participants with AEs and SAEs by treatment group, including changes in vital signs, electrocardiograms (ECGs) and laboratory results qualifying and reported as AEs.
Phase II: Number of participants with dose interruptions, reductions and discontinuations | 2 years
  Assessment of tolerability. For patients who do not tolerate the protocol-specified dosing schedule, dose adjustments are permitted in order to allow patients to continue the study treatment.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (8):
  - University of California LA, Los Angeles, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - WA Uni School Of Med, St Louis, Missouri
  - Memorial Sloan Kettering, New York, New York
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center Uni of Te, Houston, Texas
  - Fred Hutch Cancer Research, Seattle, Washington
- Australia (2):
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
- Canada (2):
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Brno, Czechia
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense C
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Saint-Herblain
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ulm
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Tel Aviv
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Chuo Ku, Tokyo, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, Korea, South Korea
- Novartis Investigative Site, Barcelona, Spain
- Novartis Investigative Site, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.